CLINICAL TRIAL: NCT06468696
Title: Improvements in Thyroid Tumor Surgery and the Prognosis, Diagnosis, Recurrence and Metastasis of Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230318
Record Dates: First submitted 2024-06-03; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Papillary Thyroid Cancer; Lymph Node Metastasis; Carcinogenesis
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis; Carcinogenesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Suturing the cervical linea alba during endoscopic thyroid surgery (Experimental): Suturing the cervical linea alba during endoscopic thyroid surgery.
  Interventions: Procedure: Suturing the cervical linea alba during endoscopic thyroid surgery.
- Not suturing the cervical linea alba during endoscopic thyroid surgery (No Intervention): Not suturing the cervical linea alba during endoscopic thyroid surgery.
- Thyroid papillary carcinoma group (Other): Thyroid papillary carcinoma tissue.
  Interventions: Genetic: Performing transcriptome sequencing
- Thyroid papillary carcinoma adjacent group (Other): Thyroid papillary carcinoma adjacent tissue.
  Interventions: Genetic: Performing transcriptome sequencing
- Lymph node metastasis group (Other): Lymph node tissue with metastasis.
  Interventions: Genetic: Performing transcriptome sequencing
- Non-lymph node metastasis group (Other): Lymph node tissue without metastasis.
  Interventions: Genetic: Performing transcriptome sequencing

INTERVENTIONS:
Procedure: Suturing the cervical linea alba during endoscopic thyroid surgery. — Suturing the cervical linea alba during endoscopic thyroid surgery.
  Arms: Suturing the cervical linea alba during endoscopic thyroid surgery
Genetic: Performing transcriptome sequencing — Performing transcriptome sequencing
  Arms: Lymph node metastasis group; Non-lymph node metastasis group; Thyroid papillary carcinoma adjacent group; Thyroid papillary carcinoma group

SUMMARY:
The objective of this research is to investigate the clinical outcomes of modified surgical techniques such as omitting the cervical linea alba suture in transthoracic endoscopic thyroidectomy. Furthermore, the study requires the collection of normal thyroid tissues, benign and malignant thyroid tumors, and lymph nodes to further clarify the mechanisms associated with the initiation, progression, metastasis, and recurrence of thyroid cancer.

DETAILED DESCRIPTION:
Study Purpose: Background and Significance Trans-axillary and trans-breast endoscopic thyroid surgery is currently the most widely used and recognized minimally invasive cosmetic thyroid surgery method. However, due to its inherent characteristics, this approach still has certain limitations that require further improvement. For example, there have been no studies reporting the short-term and long-term advantages of not suturing the cervical white line during trans-breast endoscopic thyroid surgery. Through theoretical analysis, it is suggested that not suturing the cervical white line during endoscopic thyroid surgery might be safe and feasible in terms of reducing operation time, postoperative pain, and incision complications, but this needs to be further verified.

The mechanisms underlying the occurrence, progression, metastasis, and recurrence of thyroid cancer are still not completely understood, necessitating further basic and clinically relevant research using clinical specimens.

Combining the current research progress domestically and internationally, the purpose of this study is to explore the clinical outcomes of improved surgical methods, such as not suturing the cervical white line during trans-axillary and trans-breast endoscopic thyroidectomy. In addition, the study aims to collect normal thyroid tissue, benign and malignant thyroid tumors, and lymph nodes to further elucidate the mechanisms related to the occurrence, progression, metastasis, and recurrence of thyroid cancer.

Study Procedure Before you are enrolled in the study, the doctor will conduct a detailed inquiry and record your medical history. Preoperative evaluations will include thyroid and lymph node ultrasound, neck CT, thyroid function tests, and fine-needle aspiration biopsy. If you meet the inclusion and exclusion criteria, you can voluntarily choose to participate in this study and sign an informed consent form. If you agree to participate in this study, you will be assigned a number, and a research file will be created.

This study will be conducted at the Second Affiliated Hospital of Xi'an Jiaotong University, with an estimated 200 voluntary participants. The research will involve collecting medical information data generated during routine clinical diagnosis and treatment, pathological reports, and tissue specimens from the thyroid, thyroid tumors, and lymph nodes obtained during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Perform transthoracic endoscopic thyroidectomy via breast approach;
2. Postoperative pathology confirms benign or malignant thyroid tumors;
3. Preoperative thyroid ultrasound or cervical CT suggests no extrathyroidal invasion or distant metastasis of the tumor;
4. No contraindications for general anesthesia;
5. Patients with cosmetic requirements.

Exclusion Criteria:

1. Underwent transthoracic endoscopic thyroidectomy;
2. Postoperative pathology confirmed as benign or malignant thyroid tumors;
3. Preoperative thyroid ultrasound or neck CT suggested no extraglandular invasion or distant metastasis of the tumor;
4. No contraindications to general anesthesia;
5. Patients with cosmetic demands.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative neck edema Incidence rate | Within one week post-surgery
  Postoperative neck edema Incidence rate
Postoperative short-term pain | Within one week post-surgery
  Record the patient's perception of wound pain on postoperative days 1, 3, and 5 using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst pain), for quantification.
Thyroid Papillary carcinoma tissue mRNA expression profile | Within one month after the transcriptome sequencing.
  After extracting total RNA from tissue, it is purified and a cDNA library is constructed. Following library quality control, sequencing is conducted on the Illumina NovaSeq 6000 platform using the PE150 mode to obtain tissue mRNA expression data.
Thyroid papillary carcinoma metastatic lymph node mRNA expression profile | Within one month after the transcriptome sequencing.
  After extracting total RNA from tissue, it is purified and a cDNA library is constructed. Following library quality control, sequencing is conducted on the Illumina NovaSeq 6000 platform using the PE150 mode to obtain tissue mRNA expression data.

CONTACTS AND LOCATIONS:
Overall Officials: Zhidong Wang, Principal Investigator — Xi'an Jiaotong University Second Affiliated Hospital
Locations (1):
- Xi'an Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi, China